CLINICAL TRIAL: NCT00578968
Title: Cardiac Limitations in Chronic Obstructive Pulmonary Disease: Benefits of Bronchodilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Boehringer Ingelheim (Industry); Pfizer (Industry)
Responsible Party: Bruce Johnson, PhD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-003434
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: COPD; Tiotropium; Spiriva
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tiotropium (Experimental): Participants with chronic obstructive pulmonary disease randomized to this arm received a once daily oral inhalation of 18 mcg tiotropium powder.
  Interventions: Drug: Tiotropium
- Placebo (Placebo Comparator): Participants with chronic obstructive pulmonary disease randomized to this arm received a once daily oral inhalation of placebo powder to match the standard active comparator dose.
  Interventions: Drug: Placebo
- Healthy Controls (No Intervention): Healthy age and gender matched controls were recruited for comparing cardiovascular responses to participants with chronic obstructive pulmonary disease prior to the intervention.

INTERVENTIONS:
Drug: Tiotropium — Participants received once daily Spiriva capsules for oral inhalation: 18 mcg tiotropium powder, for use with HandiHaler device.
  Other Names: Spiriva
  Arms: Tiotropium
Drug: Placebo — Participants randomized to this arm received a once daily oral inhalation of placebo powder to match the standard active comparator dose, using the HandiHaler device.
  Arms: Placebo

SUMMARY:
This study is being done to examine the influence of Tiotropium (good or bad) on heart function at rest and during exercise in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Patients who develop chronic obstructive pulmonary disease (COPD) have a loss of elastic recoil of the lungs, have remodeling in the airways and pulmonary vasculature, develop inhomogeneities in ventilation (VA) and perfusion (Qc) and gradually lose their reserves for producing expiratory flow, particularly over the mid to lower lung volumes. As a result, they develop air trapping, have slowed expiration, and gradually hyperinflate with a large residual volume, an exaggerated total lung capacity, reduced vital capacity, and markedly reduced maximal expiratory flows. With exercise, patients with moderate to severe COPD are further challenged by the need for increased ventilation. Expiring against the narrowed airways results in breathing at higher and higher lung volumes until the elastic load on inspiration increases the work and cost of breathing to the point where exercise discontinues. It remains controversial if this scenario leads to primarily dyspnea from the weak and heavily recruited inspiratory muscles, inspiratory muscle fatigue or if a primary limitation might be related to the relatively large cardiac output required for the respiratory muscles, at the expense of the locomotor muscles, resulting in leg fatigue. The expiratory load also increases intrathoracic pressure and reduces the gradient for venous return, thus having the potential to reduce cardiac output. Pulmonary hypertension develops and may influence blood flow to the left side of the heart further inhibiting cardiac output. The ineffective inspiratory pressure generation by the diaphragm may also reduce the typical benefits of the respiratory muscle pump on venous return and the marked hyperinflation may influence left ventricular filling due to competition for intrathoracic space. Thus, although COPD primarily influences the respiratory system, we believe it has profound effects on cardiac function, and during exercise this may play a particular limitation. Use of a long-acting anticholinergic agent such as Tiotropium partially reverses airway obstruction (expiratory load) and hyperinflation, both potentially improving cardiovascular function. The focus of this research will be to determine influence of Tiotropium on cardiac parameters measured both at rest and during exercise.

The focus of this study was to determine the influence of Tiotropium (Spiriva) on cardiac parameters measured both at rest and during exercise. More specifically, we first examined cardiac function in a group of COPD patients and healthy age and gender matched controls. Our hypothesis was that at rest cardiac function would be similar between groups; however, with light and heavier exercise, there would be evidence for a blunted stroke volume and perhaps cardiac output in the COPD patients. Second, we compared in a placebo-controlled double blinded manner cardiac function with and without chronic use of tiotropium in age, gender, and disease matched COPD patients. Our hypothesis was that in the Tiotropium (Spiriva) group at a matched workload, the reduced obstruction would allow for improved cardiac function, specifically an increase in stroke volume and reduction in heart rate. The interactions in this population between metabolic demand, fitness, lung mechanics, and cardiovascular function are complicated and thus studies were pursued at matched workloads and heart rate as well as with heavier exercise in an attempt to discriminate a primary influence of altered obstruction on cardiovascular function.

The participants will be asked to come to the Cardiopulmonary Research Laboratory on 4 occasions (separate visits) for exercise testing (typically over the course of 2 to 4 weeks). Each session will take approximately 1-4 hours to complete and in the COPD population, visits will be repeated after receiving placebo or Tiotropium for 4 weeks.

All of the exercise testing will be performed on an exercise bicycle either in the upright or semi-supine (recumbent) position and the participant will wear a SCUBA-type mouthpiece and a nose clip to analyze expired air. In addition, an EKG will be used to monitor heart rate and rhythm.

Visit 1 (Screening Visit): During the first visit, participants will have a brief exam by a pulmonary physician. The exam will include a complete blood count (CBC) to rule out anemia, baseline spirometry to assess lung volumes and flow rates to meet entry criteria, and in women of childbearing potential a pregnancy test. They will also be taken off theophylline and inhaled anticholinergics, but allowed to continue long acting inhaled beta agonists (LABA) or short acting beta agonist (SABA) for a rescue medication. Subjects on long acting inhaled beta agonists will be asked to discontinue this medication temporarily, 48 hr. prior to each study visit, but restarted upon completion of the visit.

Visit 2: A minimum of 48 hours after the first visit, participants will return for complete measures of lung volumes, flow rates, and diffusing capacity of the lung for carbon monoxide (DLCO), a baseline echocardiogram and a maximal exercise test on a cycle ergometer. Before the exercise begins, participants will have one or two small balloon(s) (2 inches long, deflated) attached to a small plastic tube (the width of a pencil tip) inserted through the nasal cavity and into the esophagus. This is done to measure respiratory muscle work. Participants will receive a numbing gel (2% lidocaine) to numb the nasal passage and upper esophagus prior to insertion of the balloon(s). During the insertion of the esophageal balloons, participants will also be asked to swallow water to minimize gagging and assure correct balloon placement in the esophagus. Participants will also be asked to breathe a mixture of gases containing acetylene (0.6%), dimethyl ether (1.8%), oxygen (21%, same as room air), helium (9%) and nitrogen (69.4%). The mixture of gases will be inhaled at various time points over the course of the exercise session for 8 to 10 breaths at a time. This is done to non-invasively measure cardiac output.

Visit 3: Visit 3 will involve steady-state semi-recumbent cycling exercise at two steady-state exercise intensities; 40 percent of peak work and (after a brief rest) an intensity eliciting a heart rate of 110 beats per minute (to standardize diastolic duration). Before the exercise begins, participants will have one or two small balloon(s) (2 inches long, deflated) attached to a small plastic tube (the width of a pencil tip) inserted through the nasal cavity and into the esophagus. This is done to measure respiratory muscles at work. Participants will receive a numbing gel (2% lidocaine) to numb the nasal passage and upper esophagus prior to insertion of the balloon(s). During the insertion of the esophageal balloons, participants will also be asked to swallow water to minimize gagging and assure correct balloon placement in the esophagus. Participants will also be asked to breathe a mixture of gases containing acetylene (0.6%), dimethyl ether (1.8%), oxygen (21%, same as room air), helium (9%) and nitrogen (69.4%). The mixture of gases will be inhaled at various time points over the course of the exercise session for 8 to 10 breaths at a time. This is done to non-invasively measure cardiac output. Also during the session, a sonographer will use ultrasound to measure cardiac pressures and volumes.

Visit 4: Visit 4 will involve steady-state exercise at 70% of peak work. Before the exercise begins, participants will have one or two small balloon(s) (2 inches long, deflated) attached to a small plastic tube (the width of a pencil tip) inserted through the nasal cavity and into the esophagus. This is done to measure respiratory muscles at work. Participants will receive a numbing gel (2% lidocaine) to numb the nasal passage and upper esophagus prior to insertion of the balloon(s). During the insertion of the esophageal balloons, participants will also be asked to swallow water to minimize gagging and assure correct balloon placement in the esophagus. Participants will also be asked to breathe a mixture of gases containing acetylene (0.6%), dimethyl ether (1.8%)oxygen (21%, same as room air), helium (9%) and nitrogen (69.4%). The mixture of gases will be inhaled at various time points over the course of the exercise session for 8 to 10 breaths at a time. This is done to non-invasively measure cardiac output.

Upon completion of these baseline visits, the COPD patients will be randomly assigned to a standard dose of Tiotropium once-daily (18 µg) or placebo for 4 weeks (or until study completion as visits 2-4 may require 1-2 wks to complete). Patients otherwise will receive usual care, except (as noted) for discontinuing other anticholinergic bronchodilators and theophylline. They will also discontinue long acting beta agonists for 48 hours prior to performing each of the designated visits. At the end of this intervention period, the procedures outlined in Visits 2-4 will be repeated (on the COPD patients only). All post intervention visits will be timed so that the primary measures will be made 1.5 to 2 hrs post dose of Tiotropium.

ELIGIBILITY:
Chronic obstructive pulmonary disease (COPD) participants-

Inclusion criteria:

* Body Mass Index (BMI) <36
* Moderate to severe COPD patient, (similar to or slightly better than Gold Guidelines Stage 2-3, forced expiratory volume in one second [FEV_1] <60% of age predicted)
* Smoking history of 10 pack years or more
* Clinical diagnosis of COPD
* Not on daytime oxygen

Exclusion criteria:

* Clinical diagnosis of asthma
* Myocardial infarction within the last 6 months, or known ischemia
* Serious uncontrolled cardiac arrhythmia (i.e., atrial fibrillation or ventricular tachycardia) or hospitalization for heart failure within the previous year
* Known moderate to severe renal impairment
* Known moderate to severe symptomatic prostatic hypertrophy or bladder neck obstruction
* Known narrow angle glaucoma
* Current radiation or chemotherapy for a malignant condition
* Inability to give informed consent
* On systemic corticosteroids at unstable doses or on regular daily doses of 20 mg or more of prednisone (or equivalent)
* Not fully recovered from an exacerbation of COPD for at least 30 days
* Inability to perform light to moderate activity for orthopedic reasons or who significantly desaturated with exercise (percentage of available hemoglobin that is saturated with oxygen [SaO_2] < 85% on screening test

Healthy controls -

Inclusion:

- Age and gender matched to COPD participants

Exclusion:

- Subjects who are unable to engage in exercise testing due to existing comorbidities

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Johnson, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Mayo Clinic, Rochester, Minnesota from October 2006 to August 2008. The first period compared cardiovascular response in COPD patients to healthy controls prior to the intervention. In the second period the COPD patients were randomized to drug or placebo; the controls did not take part in this period.
Period: Baseline (Prior to Intervention)
Arm/Group | Tiotropium | Placebo | Healthy Controls
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Intervention
Arm/Group | Tiotropium | Placebo | Healthy Controls
Started | 12 | 12 | 0
Completed | 12 | 12 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | Placebo | Healthy Controls | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (5.7) | 56.3 (9.4) | 58.4 (10.6) | 58.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 10
  Male | 8 | 10 | 8 | 26
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36
Height [Mean (Standard Deviation); unit: cm] | 169.1 (10.3) | 172.5 (8.0) | 173.0 (7.7) | 171.3 (8.7)
Weight [Mean (Standard Deviation); unit: kg] | 91.9 (30.2) | 89.6 (17.9) | 80.4 (11.3) | 86.7 (21.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (10.4) | 29.9 (4.4) | 26.8 (3.1) | 29.4 (7.0)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 2.06 (0.35) | 2.07 (0.25) | 1.96 (0.17) | 2.02 (0.26)

OUTCOME MEASURES:

1. Secondary Outcome: Baseline Resting Forced Vital Capacity (FVC)
Description: Vital capacity is the maximum amount of air a person can expel from the lungs after a maximum inspiration. A person's vital capacity can be measured by a spirometer which can be a wet or regular spirometer. In combination with other physiological measurements, the vital capacity can help make a diagnosis of underlying lung disease.
Time Frame: First visit of first study period
Population: All COPD participants were included, prior to randomization in the second period of the study.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- COPD Participants: All of the COPD participants were included in the first period prior to the intervention to compare cardiovascular responses to resting and exercise states with healthy controls.
- Healthy Controls: Healthy age and gender matched controls were recruited for the first period prior to the intervention to compare cardiovascular responses to resting and exercise states with COPD participants.
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
Liters | 3.29 (1.02) | 4.20 (0.98)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p = 0.01, ANOVA

2. Secondary Outcome: Baseline Resting FVC as Percentage of Predicted Forced Vital Capacity (FVC)
Description: Predicted normal values for vital capacity can be calculated online (based on previous research) and depends on age, sex, height, weight and ethnicity. Percentage was calculated by observed FVC/predicted FVC X 100.
Time Frame: First visit of first study period
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
percentage of predicted FVC | 78.3 (13.8) | 99.4 (14.8)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Baseline Resting Forced Expiratory Volume in 1 Second (FEV_1)
Description: FEV_1 is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity.
Time Frame: first visit of first study period
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
L/sec | 1.74 (0.70) | 3.22 (0.74)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p < 0.001, ANOVA

4. Secondary Outcome: Baseline Resting FEV_1 as Percentage of Predicted FEV_1
Description: Predicted normal values for Forced Expiratory Volume in 1 second can be calculated online (based on previous research) and depends on age, sex, height, weight and ethnicity. Percentage was calculated by observed FEV_1/predicted FEV_1 X 100.
Time Frame: first visit of first study period
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV_1
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
percentage of predicted FEV_1 | 51.6 (14.1) | 97.5 (12.4)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p < 0.001, ANOVA

5. Secondary Outcome: Baseline Heart Rate (HR) for All COPD Participants Versus Healthy Control Groups
Description: Heart rate is the number of heartbeats per unit of time, typically expressed as beats per minute (bpm). Heart rate was measured in the first study period prior to the intervention at resting and at peak exercise states.
Time Frame: first visit of first study period, second visit of first study period
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
beats per minute (bpm)
  Baseline Resting, V1-1st study period | 79.4 (13.7) | 72.7 (10.4)
  Baseline Peak Exercise, V2-1st study period | 127.8 (23.4) | 153.6 (16.8)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Comparison between the two groups at baseline resting; Test type: Superiority or Other; p = 0.13, ANOVA
Statistical Analysis 2: Comparison: COPD Participants vs Healthy Controls; Comparison was made between the two groups at baseline peak exercise; Test type: Superiority or Other; p < 0.01, ANOVA

6. Secondary Outcome: Baseline Peak Exercise Maximal Oxygen Consumption (VO_2)
Description: VO_2 is the maximum capacity of an individual's body to transport and use oxygen during incremental exercise.
Time Frame: second visit of first study period
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
L/min | 1.52 (0.41) | 2.29 (0.60)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p < 0.001, ANOVA

7. Secondary Outcome: Baseline Peak Exercise Cardiac Index (CI)
Description: Cardiac index: A cardiodynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area (m^2) to yield the cardiac index.
Time Frame: second visit of first study period
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
L/min/m^2 | 6.02 (1.65) | 7.61 (2.14)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p < 0.05, ANOVA

8. Secondary Outcome: Baseline Peak Exercise Stroke Volume Index (SVI)
Description: Stroke volume - the volume of blood ejected from a ventricle at each beat of the heart, equal to the difference between the end-diastolic volume and the end-systolic volume. The stroke volume index is a method of relating the stroke volume to the size of the person by dividing the stroke volume by the BSA (m^2).
Time Frame: second visit of first study period
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
mL/m^2 | 47.3 (11.0) | 52.7 (9.4)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p = 0.15, ANOVA

9. Secondary Outcome: Pretreatment Resting Forced Vital Capacity (FVC)
Description: as for outcome 1
Time Frame: First study visit of first study period
Population: Normal Control population did not take part in this measurement. Researchers collected this data V1 study period 1, but randomized subjects after V4 study period 1.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
Liters | 2.79 (0.64) | 3.80 (1.10)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.01, ANOVA

10. Primary Outcome: Baseline Resting Cardiac Index (CI)
Description: as for outcome 7
Time Frame: First visit of first study period
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
L/min/m^2 | 2.4 (0.71) | 2.36 (0.51)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p = 0.85, ANOVA

11. Primary Outcome: Baseline Resting Stroke Volume Index (SVI)
Description: Stroke volume - the volume of blood ejected from a ventricle at each beat of the heart, equal to the difference between the end-diastolic volume and the end-systolic volume. The stroke volume index is a method of relating the stroke volume to the size of the person by dividing the stroke volume by the body surface area (BSA) (m^2).
Time Frame: first visit of first study period
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | COPD Participants | Healthy Controls
Number analyzed (Participants) | 24 | 12
mL/m^2 | 31.3 (11.5) | 39.7 (8.3)
Statistical Analysis 1: Comparison: COPD Participants vs Healthy Controls; Test type: Superiority or Other; p = 0.03, ANOVA

12. Secondary Outcome: Pretreatment Resting FVC as Percentage of Predicted FVC
Description: as for outcome 2
Time Frame: First visit of first period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
percentage of predicted FVC | 71.24 (9.08) | 85.27 (14.34)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.009, ANOVA

13. Secondary Outcome: Percent Change in Resting FVC Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: Vital capacity is the maximum amount of air a person can expel from the lungs after a maximum inspiration. A person's vital capacity can be measured by a spirometer which can be a wet or regular spirometer. In combination with other physiological measurements, the vital capacity can help make a diagnosis of underlying lung disease. Percentage change = final value - initial value/initial value x 100
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal Control population did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: percentage of change in FVC
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
percentage of change in FVC | 11.55 (15.27) | -6.20 (11.03)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.005, ANOVA

14. Secondary Outcome: Pretreatment Resting FEV_1
Description: as for outcome 3
Time Frame: first study visit of first study period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
L/sec | 1.48 (0.49) | 2.00 (0.80)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.06, ANOVA

15. Secondary Outcome: Percent Change in Resting FEV_1 Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: FEV_1 is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. Percentage change = final value - initial value/initial value x 100
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal controls did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: Percentage of change in FEV_1
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
Percentage of change in FEV_1 | 8.81 (11.86) | -6.30 (1.98)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.003, ANOVA

16. Secondary Outcome: Pretreatment Resting CI
Description: Cardiac index (CI): A cardiodynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area (m^2) to yield the cardiac index.
Time Frame: first study visit of first study period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
L/min/m^2 | 2.31 (0.72) | 2.49 (0.73)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.60, ANOVA

17. Secondary Outcome: Percent Change in Resting CI Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: Cardiac index (CI): A cardiodynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area (m^2) to yield the cardiac index. Percentage change = final value - initial value/initial value x 100
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal controls did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: percentage of change in CI
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
percentage of change in CI | -4.91 (26.80) | -9.08 (25.04)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.35, ANOVA

18. Secondary Outcome: Pretreatment Resting SVI
Description: as for outcome 8
Time Frame: first study visit of first study period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
mL/m^2 | 30.08 (12.59) | 32.55 (10.69)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.65, ANOVA

19. Secondary Outcome: Percent Change in Resting SVI Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: Stroke volume - the volume of blood ejected from a ventricle at each beat of the heart, equal to the difference between the end-diastolic volume and the end-systolic volume. The stroke volume index is a method of relating the stroke volume to the size of the person by dividing the stroke volume by the BSA (m^2). Percentage change = final value - initial value/initial value x 100
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal controls did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: Percentage of change in SVI
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
Percentage of change in SVI | -3.80 (34.54) | -6.26 (29.15)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.43, ANOVA

20. Secondary Outcome: Pretreatment Heart Rate (HR) in Tiotropium and Placebo Groups
Description: as for outcome 5
Time Frame: first study visit of first study period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
bpm
  Pretreatment Resting HR, V1-1st study period | 80.50 (15.37) | 78.33 (12.32)
  Pretreatment Peak Exercise HR, V1-1st study period | 120.17 (21.44) | 135.33 (23.67)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Comparison was made between groups at pretreatment resting time period; Test type: Superiority or Other; p = 0.73, ANOVA
Statistical Analysis 2: Comparison: Tiotropium vs Placebo; Comparison was made between groups at pretreatment peak exercise time period; Test type: Superiority or Other; p = 0.11, ANOVA

21. Secondary Outcome: Percent Change in Resting HR Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: Heart rate is the number of heartbeats per unit of time, typically expressed as beats per minute (bpm). Percentage change = final value - initial value/initial value x 100
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal control population did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: Percentage of change in HR
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
Percentage of change in HR | -7.05 (5.14) | -1.32 (8.35)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.22, ANOVA

22. Secondary Outcome: Pretreatment Peak Exercise Maximal Oxygen Consumption (VO_2)
Description: VO_2 is the maximum capacity of an individual's body to transport and use oxygen during incremental exercise.
Time Frame: first visit of first study period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
L/min | 1.33 (0.33) | 1.65 (0.46)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.06, ANOVA

23. Secondary Outcome: Percent Change in Peak Exercise VO_2 Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: VO_2 is the maximum capacity of an individual's body to transport and use oxygen during incremental exercise. Percentage change = final value - initial value/initial value x 100
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal Control population did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: percentage of change in VO_2
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
percentage of change in VO_2 | 2.06 (12.76) | -4.60 (10.27)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.09, ANOVA

24. Primary Outcome: Pretreatment Peak Exercise CI
Description: as for outcome 16
Time Frame: first visit of first study period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
L/min/m^2 | 5.34 (1.39) | 6.70 (1.66)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.04, ANOVA

25. Secondary Outcome: Percent Change in Peak Exercise CI Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: as for outcome 17
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal control population did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: percentage of change in CI
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
percentage of change in CI | 2.46 (14.02) | -11.80 (21.29)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.04, ANOVA

26. Primary Outcome: Pretreatment Peak Exercise SVI
Description: as for outcome 8
Time Frame: first visit of first study period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
mL/m^2 | 44.62 (9.0) | 50.06 (12.49)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.19, ANOVA

27. Secondary Outcome: Percent Change in Peak Exercise SVI Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: as for outcome 19
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal control population did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: percentage of change in SVI
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
percentage of change in SVI | 3.11 (16.37) | -4.95 (21.33)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.16, ANOVA

28. Secondary Outcome: Percent Change in Peak Exercise HR Between Pretreatment in First Study Period and Post-treatment in Second Study Period
Description: as for outcome 21
Time Frame: first visit of first study period, first visit of second study period (approximately 6 weeks later)
Population: Normal control population did not take part in this measurement.
Measure: Mean (Standard Deviation); unit: percentage of change in HR
Arm/Group | Tiotropium | Placebo
Number analyzed (Participants) | 12 | 12
percentage of change in HR | 0.27 (12.30) | -7.05 (5.14)
Statistical Analysis 1: Comparison: Tiotropium vs Placebo; Test type: Superiority or Other; p = 0.04, ANOVA

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events from baseline through the last study visit, approximately 12 weeks.
Arm/Group | Tiotropium | Placebo | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No